CLINICAL TRIAL: NCT05803642
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Injection of Olanzapine in the Treatment of Acute Agitation Associated With Schizophrenia and Bipolar I Disorder.
Brief Title: A Study of Olanzapine in Patients With Acute Agitation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QLG2072-301
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Acute Agitation
MeSH Terms: interventions — Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine (Experimental)
  Interventions: Drug: Olanzapine
- Haloperidol (Active Comparator)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Olanzapine — intramuscular injection, 10 mg/dose, first dose and an optional second or third dose.
  Arms: Olanzapine
Drug: Haloperidol — intramuscular injection, 7.5 mg/dose, first dose and an optional second or third dose.
  Arms: Haloperidol

SUMMARY:
The purpose of this study is to assess the efficacy and safety of intramuscular olanzapine for the treatment of acute agitation associated with schizophrenia and bipolar I mania.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 to 65 years, inclusive.
2. Patients who have met DSM-5 criteria for schizophrenia and bipolar I disorder.
3. Patients who are judged to be clinically acutely agitated with a total score of ≥ 14 on the 5 items comprising the PANSS-EC and at least one individual item score≥ 4 immediately before randomization.

Exclusion Criteria:

1. Patients with agitation caused by delirium, seizures, developmental delay, poisoning, etc., or withdrawal from drug abuse.
2. Patients who have had previous suicidal behavior or currently at serious risk of suicide.
3. Patients with glaucoma or at risk of angle-closure glaucoma.
4. Patients who have brain diseases such as intracranial infection, brain trauma, cerebrovascular disease, basal ganglion disease, hypoxic encephalopathy, Parkinson's disease, Parkinson's syndrome, and dementia.
5. Use of benzodiazepines, other hypnotics or short-acting antipsychotic drugs within 4 hours before randomization.
6. Treatment with psychostimulants or reserpine within one week before randomization.
7. Patients who received long-acting injections of typical or atypical antipsychotics within 2 weeks prior to randomization or within one injection interval.
8. Treatment with clozapine within 4 weeks before screening.
9. Patients with serious or unstable medical illnesses.
10. Female patients who have a positive pregnancy test at screening or are breastfeeding.
11. Patients who have participated in other clinical trials within 3 months before randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-03-28 (Estimated); Primary Completion 2024-05-07 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 2 hours post-first IM injection on the PANSS-EC | 2 hours
  The PANSS-EC comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)

SECONDARY OUTCOMES:
Percentage of Participants With 40% or Greater Percent Decrease in the PANSS-EC Total Score | 2 hours post-first IM injection
Proportion of participants receiving one, two, or three doses of study drug during 24-hour intramuscular treatment period | 24 hours